CLINICAL TRIAL: NCT00884806
Title: Corneal Staining Evaluation of SiH MPDS FID 114675A
Brief Title: 7-Day, Multi-Site Study of an Investigational Multi-Purpose Disinfecting Solution for Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C-08-081
Record Dates: First submitted 2009-04-17; First posted 2009-04-21 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Contact Lens Care
Keywords: Contact lenses; Disinfecting solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 114675A (Experimental): FID 114675A used for 7 days, per protocol-specified instructions. Silicone hydrogel or hydrogel contact lenses worn bilaterally on a daily wear basis, one brand only.
  Interventions: Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS); Device: Etafilcon A contact lens (ACUVUE® 2™); Device: Senofilcon A contact lens (ACUVUE® OASYS™); Device: Lotrafilcon B contact lens (O2 OPTIX®); Device: Balafilcon A contact lens (PureVision®)

INTERVENTIONS:
Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS) — Investigational solution intended for use as a cleaning, rinsing, conditioning, disinfecting, and storage solution for silicone hydrogel (SiH) contact lenses
Device: Etafilcon A contact lens (ACUVUE® 2™) — Commercially marketed hydrogel contact lens for daily wear use
  Other Names: ACUVUE® 2™
Device: Senofilcon A contact lens (ACUVUE® OASYS™) — Commercially marketed silicone hydrogel contact lens for daily wear use
  Other Names: ACUVUE® OASYS™
Device: Lotrafilcon B contact lens (O2 OPTIX®) — Commercially marketed silicone hydrogel contact lens for daily wear use
  Other Names: O2 OPTIX®
Device: Balafilcon A contact lens (PureVision®) — Commercially marketed silicone hydrogel contact lens for daily wear use
  Other Names: PureVision®

SUMMARY:
The purpose of this study is to clinically evaluate solution-related corneal staining with an investigational multi-purpose disinfecting solution (MPDS) in hydrogel and silicone hydrogel contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Wear contact lenses a minimum of 8 hours per day for at least 7-10 days prior to Visit 1 (screening visit).
* Vision correctable to 20/30 (Snellen) or better in each eye at distance with contact lenses at Visit 1.
* Must discontinue contact lens wear for at least two consecutive days before Visit 2 (baseline visit).
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any medical condition (systemic or ophthalmic) that may, in the opinion of the investigator, preclude safe administration of test article or safe participation in the study.
* Known sensitivity or intolerance to any protocol-specified contact lens solutions, eye drops, or products containing similar ingredients (e.g., generic products).
* Monocular vision (only one eye with functional vision) or fit with only one contact lens.
* Use of topical ocular over-the-counter or prescribed topical ocular medication, with the exception of rewetting drops, within 7 days prior to screening visit.
* Current or history of ocular infection, inflammation, disease, structural abnormality or conditions within the last 6 months that could affect study participation or may preclude safe administration of the investigational lens care solution, in the opinion of the investigator.
* Any corneal surgery, cataract surgery, intraocular lens implants or glaucoma filtering surgery within the last 12 months.
* Any slit-lamp finding score of 1 (or rated 3 or 4 for limbal and bulbar conjunctival injection) at screening or baseline visits.
* Corneal staining area assessment ≥ 20% in any corneal region in either eye at baseline visit.
* Corneal staining graded as 2 (macropunctate) or greater in any corneal region in either eye at baseline visit.
* Participation in any investigational clinical study within 30 days of baseline visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 US study centers.
Pre-assignment Details: 110 participants with normal eyes (other than vision correction) were enrolled in the study. After the screening visit, particpants discontinued contact lens wear and wore their glasses for at least 2 days as a washout prior to the baseline/dispensing visit.
Groups:
- FID 114675A: FID 114675A used 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel or hydrogel contact lenses, per protocol-specified instructions.
Period: Overall Study
Arm/Group | FID 114675A
Started | 110
Completed | 110
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FID 114675A
Number analyzed (Participants) | 110
Age Continuous [Mean (Standard Deviation); unit: years] | 33.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Solution-Related Corneal Staining
Description: Corneal staining was assessed by the investigator using fluorescein dye, a yellow filter, and a slit lamp. Corneal staining was graded on a continuous scale of 0% (no staining in the region) to 100% (staining covers entire region) in 1% increments for 5 corneal regions (central, nasal, temporal, inferior, and superior). Solution-related corneal staining was defined as ≥20% corneal staining area in at least 3 corneal regions of both eyes.
Time Frame: Day 7
Population: Intent to treat: All participants who received regimen and had at least one on-therapy visit.
Measure: Number; unit: Percentage of participants
Arm/Group | FID 114675A
Number analyzed (Participants) | 110
Percentage of participants | 0

2. Secondary Outcome: Mean Lens Comfort
Description: Lens comfort was assessed by the participant on a 5-point Likert scale prior to any examination. The participant was instructed to select a single response to the statement, "Over the previous 2-3 hours, my lenses felt comfortable," with 1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, and 5 = strongly agree.
Time Frame: Day 7
Population: Intent to treat: All participant who received regimen and had at least one on-therapy study visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FID 114675A
Number analyzed (Participants) | 28
Units on a scale | 4.4 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 24 March 2009 to 19 June 2009.
Description: This reporting group includes all participants enrolled and exposed to test regimen.
Groups:
- FID 114675A: Investigational multi-purpose contact lens solution
Arm/Group | FID 114675A
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.